CLINICAL TRIAL: NCT03693716
Title: Arthroscopic Dynamic Anterior Capsular Stabilization With Trans Subscapular Long Head of the Biceps Tenodesis in Anterior Shoulder Instability - Clinical and Imagiological Results
Brief Title: Dynamic Anterior Stabilization With Transsubscapular Long Head of the Biceps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Egas Moniz (Other)
Collaborators: Centro Hospitalar Lisboa Ocidental (Other Government)
Responsible Party: Principal Investigator, Clara Isabel de Campos Azevedo, Shoulder Surgery Unit Coordinator, Hospital de Egas Moniz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-2018-09HSFX
Record Dates: First submitted 2018-09-30; First posted 2018-10-03 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Anterior Shoulder Dislocation; Bankart Lesion; Hill Sachs Lesion
Keywords: Transsubscapular; Long head of the biceps tendon; LHBT; Anterior Shoulder Dislocation; Bankart; HillSachs; Arthroscopic Anterior Dynamic Stabilization
MeSH Terms: conditions — Bankart Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dynamic Anterior Stabilization (Experimental): Arthroscopic Dynamic Anterior Capsular Stabilization with Trans subscapular Long Head of the Biceps Tenodesis
  Interventions: Procedure: Dynamic Anterior Stabilization

INTERVENTIONS:
Procedure: Dynamic Anterior Stabilization — All-arthroscopic trans subscapular Long Head of the Biceps tenodesis in the anterior-inferior glenoid with all-suture anchors

SUMMARY:
Clinical study of patients with a history of traumatic anterior shoulder dislocations to test the hypothesis that the arthroscopic dynamic anterior capsular stabilization technique with trans subscapular long head of the biceps tenodesis produces progressive good clinical and imagiological results.

DETAILED DESCRIPTION:
Patients with a history of traumatic anterior shoulder dislocations with documented imagological Bankart and HillSachs lesions who meet the eligibility criteria will be enrolled in the study and undergo an arthroscopic dynamic anterior capsular stabilization technique with trans subscapular long head of the biceps tenodesis. All patients will be clinically and radiologically/imagiologically assessed preoperatively and at the 6-months, 12-months and 2-years postoperative evaluations. The range of motion (ROM), shoulder abduction strength, Constant, ROWE and WOSI scores will be compared from preoperative to 6 months postoperative; from 6 months postoperative to 12 months postoperative; and from 12 months to 2 years postoperative (paired-samples t-test, two-tailed). All continuous variables will be compared between the group of patients with failures (a failure is defined as a patient who suffers an objective re-dislocation episode during the 2-year follow-up) and the group without failures (Mann-Whitney U test). All categorical variables and outcome results will be compared between the two groups (Fisher's exact test). A significant difference will be defined as P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Bankart lesion and Hill Sachs lesions on the magnetic resonance imaging
* one or more traumatic anterior shoulder dislocation episodes
* contact or forced overhead sport or work activity

Exclusion Criteria:

* proximal humerus fracture
* rotator cuff tear requiring repair

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Shoulder range of motion (ROM) | 2 years
  Bilateral shoulder active range of motion (ROM): elevation (0 -180º), abduction (0 -180º) and external rotation (0 -100º), measured in degrees ; and internal rotation, defined as the highest vertebral body that the patient's thumb can reach, converted afterwards to a scale of 1-5 points: lateral thigh=0; buttock=1; sacrum=2; lumbar=3; 12th thoracic vertebra=4; 7th thoracic vertebra=5; for every scale range provided, higher values represent a better outcome.

SECONDARY OUTCOMES:
Shoulder Strength | 2 years
  minimum 0 - maximum 25 kilograms, measured using a digital dynamometer; for every scale range provided, higher values represent a better outcome.
The ROWE score | 2 years
  0 -100 points: Section 1 - Stability No Recurrence, subluxation or apprehension (50 points) Apprehension when placing arm in certain positions (30 points) Subluxation (not requiring reduction) (10 points) Recurrent Dislocation (0 points)
  Section 2 - Motion 100% of normal ext rotation, int rotation and elevation (20 points) 75% of normal ext rotation, int rotation and elevation (15 points) 50% of normal ext rotation, int rotation and elevation (5 points) 50% of normal elevation, and int rotation, No ext rotation (0 points)
  Section 3 - Function No limitation of work or sports, little or no discomfort (eg shoulder strong overhead, lifting, swimming, throwing, tennis) (30 points)
  Mild limitation and minimum discomfort (25 points) Moderate limitation and discomfort (10 points) Marked limitation and pain (0 points) For every scale range provided, higher values represent a better outcome.
The Western Ontario Shoulder Instability Index (WOSI) | 2 years
  0-2100 (0-100%), the WOSI score instrument (Kirkley et al. 1998) consists of 21 items. The patient is asked to grade the function of a specific item on a horizontal visual analog scale from 0 to 100; for every scale range provided, higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Clara Azevedo, MD, Principal Investigator — Centro Hospitalar de Lisboa Ocidental
Locations (1):
- Centro Hospitalar de Lisboa Ocidental, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rowe CR, Patel D, Southmayd WW. The Bankart procedure: a long-term end-result study. J Bone Joint Surg Am. 1978 Jan;60(1):1-16. PMID 624747
- [Result] Kirkley A, Griffin S, McLintock H, Ng L. The development and evaluation of a disease-specific quality of life measurement tool for shoulder instability. The Western Ontario Shoulder Instability Index (WOSI). Am J Sports Med. 1998 Nov-Dec;26(6):764-72. doi: 10.1177/03635465980260060501. PMID 9850776
- [Derived] de Campos Azevedo C, Angelo AC. All-Suture Anchor Dynamic Anterior Stabilization Produced Successful Healing of the Biceps Tendon: A Report of 3 Cases. JBJS Case Connect. 2021 Feb 17;11(1). doi: 10.2106/JBJS.CC.20.00149. PMID 33599463